CLINICAL TRIAL: NCT01563458
Title: A Multi-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Dose Exploratory Trial Evaluating the Safety and Efficacy of Activated Recombinant Factor VII (rFVIIa/NovoSeven®) in the Reduction of Bleeding in Subjects Undergoing Orthotopic Liver Transplantation
Brief Title: Safety and Efficacy of Activated Recombinant Human Factor VII in Patients Undergoing Orthotopic Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7LIVER-1256
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Bleeding During/Following Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High dose (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Low dose (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — 120 mcg/kg into the vein (i.v.) bolus injection first administered immediately prior to first skin cut. Repeated every two hours until approx. 30 minutes prior to expected start of the reperfusion of the transplanted liver. 120 mcg/kg single bolus administration at completion of wound closure
  Arms: High dose
Drug: activated recombinant human factor VII — 60 mcg/kg into the vein (i.v.) bolus injection first administered immediately prior to first skin cut. Repeated every two hours until approx. 30 minutes prior to expected start of the reperfusion of the transplanted liver. 60 mcg/kg single bolus administration at completion of wound closure
  Arms: Low dose
Drug: placebo — Trial drug into the vein (i.v.) bolus injection first administered immediately prior to first skin cut. Repeated every two hours until approx. 30 minutes prior to expected start of the reperfusion of the transplanted liver. Single bolus administration at completion of wound closure
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe, North America and Oceania. The aim of this trial is to evaluate the haemostatic efficacy of activated recombinant human factor VII in subjects undergoing orthotopic liver transplantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo orthotopic liver transplantation
* Liver disease classified as Child-Turcotte (Pughs modification) score B or C

Exclusion Criteria:

* Previous liver transplantation
* Scheduled multi-organ transplantation
* Scheduled for living related donor transplantation
* Present renal insufficiency requiring dialysis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2001-08; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Total number of RBC units transfused during the perioperative period

SECONDARY OUTCOMES:
Number of RBC units transfused by surgical phase
Adverse events
Changes in coagulation related parameters

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (18):
- Australia (2):
  - Novo Nordisk Investigational Site, Camperdown
  - Novo Nordisk Investigational Site, Heidelberg
- Canada (4):
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Québec
  - Novo Nordisk Investigational Site, Toronto
- Novo Nordisk Investigational Site, Clichy, France
- Germany (2):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Essen
- Spain (3):
  - Novo Nordisk Investigational Site, Barakaldo
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Valencia
- Sweden (2):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Stockholm
- United Kingdom (4):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, London

REFERENCES:
- [Result] Lodge JP, Jonas S, Jones RM, Olausson M, Mir-Pallardo J, Soefelt S, Garcia-Valdecasas JC, McAlister V, Mirza DF; rFVIIa OLT Study Group. Efficacy and safety of repeated perioperative doses of recombinant factor VIIa in liver transplantation. Liver Transpl. 2005 Aug;11(8):973-9. doi: 10.1002/lt.20470. PMID 16035095
- [Result] Levy JH, Fingerhut A, Brott T, Langbakke IH, Erhardtsen E, Porte RJ. Recombinant factor VIIa in patients with coagulopathy secondary to anticoagulant therapy, cirrhosis, or severe traumatic injury: review of safety profile. Transfusion. 2006 Jun;46(6):919-33. doi: 10.1111/j.1537-2995.2006.00824.x. PMID 16734808
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com